CLINICAL TRIAL: NCT04452682
Title: The Impact of COVID-19 Pandemic on Critical Limb Threatening Ischemia and Emergency Vascular Practice
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R.20.06.898 - 2020/06/16
Record Dates: First submitted 2020-06-21; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: COVID; Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Era of COVID 19: Total number of cases admitted during first six months of 2020
  Interventions: Other: COVID 19 impact
- Era of Non COVID 19: Total number of cases admitted the first six months of 2019

INTERVENTIONS:
Other: COVID 19 impact — The impact of COVID-19 pandemic on Critical limb threatening ischemia and emergency vascular practice
  Groups: Era of COVID 19

SUMMARY:
This is a retrospective analytical study conducted at Vascular and Endovascular surgery Department, Mansoura University Hospital, including all patients admitted at the two periods first six months of 2019 and 2020.To demonstrate the effect of COVID-19 pandemic on the practice of emergency vascular surgery and critical limb threatening ischemia interventions by comparison two periods first six months of 2019 and 2020.

DETAILED DESCRIPTION:
INTRODUCTION:

The novel coronavirus pneumonia (COVID-19) pandemic has affected the globe, with Italy leading many reports of the incidence and mortalities. Recently reported studies have described the clinical characteristics and overall outcomes of patients with COVID-19 and the effects of treating these patients on the healthcare system.Two studies have reported associated coagulopathy disorders. These reports have highlighted the presence of a coexisting hypercoagulable state in patients with COVID-19, which might be associated with higher mortality.

The COVID-19 pandemic has had many impacts, both seen and unforeseen, all over the world. As expected, elective endovascular procedures have been halted, with a significant decrease in urgent/emergent procedures. This could reflect an understandable unwillingness on the part of patients who continue to self-isolate at home to come in for treatments, including those with Critical limb threatening ischemia. Also impacts on the supply chain side of performing interventions, had been reported, it is challenging to be in the middle of a complex CLTI (Critical limb threatening ischemia) case and request a routine device only to find out it is unavailable.

Aim of the work Evaluation the impact of COVID-19 pandemic on emergency vascular practice and critical limb ischemia.

Outcome

Primary outcomes:

* Frequencies of patients admitted at the Vascular.
* Predisposing Factors.
* Number of ICU admission.

Secondary outcomes:

• Mortality rates

Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura university hospitals Type of study: Observational analytical study Study duration: 2019-2020 Sample size: It will include all patients presented to our department at the first 6 months of 2019 and first 6 months of 2020. sample size will be 140-400 patients Inclusion criteria: all patients admitted to our department at that periods Exclusion criteria

1. Patients can't give consent (unconscious).
2. Those with mental or behavioral disorders will be excluded. Consent: Patients after signing informed consent that possible complication from the procedure ought to happen and what are the alternatives.

Data collection:

* All patients with complete medical records available will be documented
* Each patient's record will be analyzed to determine preexisting illnesses, admitting symptoms (including length of time to accessing medical care), admission physical findings, laboratory and results.
* Also, the type and duration of antibiotic therapy, the frequency and type of operative procedures performed and subsequent complications.
* Supporting modalities such as dialysis, blood product transfusion, and mechanical ventilation will be were reviewed.
* Each patient's premorbid medical profile, condition at admission, and subsequent treatment also will be analyzed to assess effect on mortality and development of complications.
* Standard treatment after admission including cardiovascular stabilization and assessment of extent of infection. Broad-spectrum antibiotics were administered to cover gram-positive cocci, gram-negative enteric rods, and anaerobic flora will be also reported.
* The procedure of Surgical Management will be described.

Statistical analysis

· The data will be analyzed using Statistical Package for the Social Sciences. The numerical outcomes e.g. age is calculated as median. Gender will be recorded as frequency and percentage. Chi Square test is applied to assess the association of various parameters. The results will be considered statistically significant if the p-value is found to be less than or equal to 0.05. To assess possible risk factors for mortality, univariate analyses will be completed initially to aid in determining the variables that should be included in a stepwise logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to our department at that periods.

Exclusion Criteria:

* Patients can't give consent (unconscious).
* Those with mental or behavioral disorders will be excluded.

Age Groups: Child, Adult, Older Adult
Study Population: It will include all patients presented to our department at the first 6 months of 2019 and first 6 months of 2020.
Sampling Method: Non-Probability Sample
Enrollment: 998 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-06-21 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
The ICU admission with associated Pneumonia | 6 months
  The ICU admission caused by Pneumonia proved radio-logically at both periods
Impact of COVID-19 on the different presentation of vascular surgery at the emergency | 6 months
  percentage of different diagnoses at both periods

SECONDARY OUTCOMES:
Mortality rates | 6 months
  Mortality percentages at both periods

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No